CLINICAL TRIAL: NCT04222153
Title: Approccio Innovativo di Trapianto di Microbiota Fecale Applicato Alla Malattia Renale Cronica
Brief Title: Innovative Approach to Fecal Microbiota Transplantation (FMT) Applied for Chronic Kidney Disease (CKD)
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Bari Aldo Moro (Other)
Responsible Party: Sponsor
Other Study IDs: FMT01
Record Dates: First submitted 2019-12-04; First posted 2020-01-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Chronic Kidney Diseases
Keywords: Fecal Microbiota Transplantation (FMT); Gut microbiota; Uremic toxins
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this PhD project focuses on the relationship between intestinal microbiota and health in the background of Chronic Kidney Disease (CKD). Many pathologies, including the CKD, display a dysbiosis of the intestinal microbiota, which is at the same time a consequence of CKD and contributes to its progression and complication. In a variety of chronic-degenerative and infectious diseases, the "fecal microbiota transplantation" (FMT) is being tested in recent years in addition with the application of both probiotics and prebiotics. FMT is indeed currently successfully used in the eradication of recurrent Clostridium difficile infections, with success rates of 90%, thus recent evidence suggests that FMT could be applied in other diseases characterized by microbiota dysbiosis, such as CKD and diabetes, in which the FMT has never been previously tested.

This project will allow to study:

i) the prototypal production of the encapsulated suspension of healthy microbiota tested in a minimally invasive FMT procedure (by oral administration);

ii) the efficacy of the innovative prototype for colonization and modulation of intestinal microbiota following FMT;

iii) the experimental and clinical feedback of this suspension, by in vivo studies.

DETAILED DESCRIPTION:
This project will allow to experiment the Fecal microbiota transplantation in the CKD model and to set up a pharmaceutical formulation of fecal suspensions of microbiota.

Firstly, a collection of fecal samples from healthy volunteers will be set up, with the aim to collect biological samples. Screening and enrollment of healthy volunteers, gathering personal and clinical information together with eating habits, will be performed.

The best product design in efficacy, stability over time as well as suitable excipients and any other active components able to perform a synergistic action will be evaluated. After defining the pharmaceutical formulation, the production of the prototype will be finalized.

In a second time in vivo studies on a model of CKD (uremic mouse with CKD induced by 5/6 nephrectomy) will be designed and carried on. The CKD model will be used to evaluate the effects and the outcomes of FMT on clinical parameters such as renal function, circulating levels of uremic toxins, state and function of the intestinal microbiota, intestinal permeability and microbiota composition. This step will be necessary to establish the efficacy of the innovative prototype for the colonization and the modulation of intestinal microbiota following FMT.

ELIGIBILITY:
Criteria: Healthy volunteers

Inclusion Criteria:

* Healthy subjects
* Aged between 18 and 50
* BMI between 18.5-25
* Omnivorous diet
* Informed consent signed

Exclusion Criteria:

* Health workers (to exclude the risk of transmission of multi-resistant organisms)
* Type 2 diabetes mellitus
* Hypertension
* Chronic liver disease
* Chronic gastrointestinal disorders
* Systemic inflammatory disorders
* Suspected, clinical diagnosis or previous history of malignancies (<5 years)
* Therapies with corticosteroids or immunosuppressive drugs
* Autoimmune disorders
* Previous history of organ / tissue transplantation
* Prior gastrointestinal surgery (eg gastric bypass)
* eGFR lower than 60ml / minute and / or diagnosis of nephropathy
* Previous acute major cardiovascular diseases (myocardial infarction, stroke)
* History of C. difficile infections
* Known systemic infection not controlled
* Previous use of antibiotics (<3 months)
* Recent appearance of diarrhea
* Chronic use of laxatives or chronic diarrhea
* Chronic constipation
* Recurrent urinary tract infections (3 cases per year)
* Use of proton pump inhibitors in the last 3 months
* Recent use of probiotics or other aids (drugs / supplements) for the regulation of gastrointestinal activity (<3 months)
* Pregnancy and breastfeeding
* Psychiatric conditions that reduce compliance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed by healthy volunteers, aged between 18 and 50, with normal BMI and characterized by omnivorous diet.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
Number of healthy volunteers enrolled according to the procedures of the FMT01 protocol | 2 months
  A final number of 10 healthy volunteers will be selected to collect their fecal samples, according to the protocol FMT01 (ref. Cammarota G et al. Gut 2017 doi:10.1136/gutjnl-2016-313017):
  1. Preliminary interview - anamnestic interview to exclude people with history of disease and risk factors
  2. Secondary interview - anamnestic interview (on the day of donation) to exclude donors with recently appeared harmful issues
  3. Sample collection - blood and stool testing to verify the presence of potentially transmittable disease: Cytomegalovirus, Epstein-Barr virus, Hepatitis A, HBV, HCV, Syphilis, HIV-1 and HIV-2, Faecal Helicobacter pylori, Faecal occult blood testing, Fecal ova and parasites Steps 1 and 2 will be analyzed by the physician in order to exclude people, after enrollment, at risk of potential harmful issues. People passing steps 1 and 2 will undergo blood and fecal laboratory screening. Positivity to one or more of the tested factor will result in volunteer exclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, MD Full Prof, Principal Investigator — Nephrology, Dialysis and Transplantation Unit "Aldo Moro" University of Bari
Locations (1):
- AUO Policlinico Consorziale, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided